CLINICAL TRIAL: NCT05665322
Title: Translate Title: Evaluation of the Efficacy of Two Guidance Techniques (Standard Injected CT vs Porto-scanner With Angio-CT) for Thermoablation Treatment of Colorectal Cancer Liver Metastases: Randomized, Single-blind, Controlled Study
Brief Title: Evaluation of the Efficacy of Two Guidance Techniques (Standard Injected CT vs Porto-scanner With Angio-CT) for Thermoablation Treatment of Colorectal Cancer Liver Metastases
Acronym: MARGIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Not enough inclusions
  * Montpellier is not included (0 inclusions)
  * Of the 7 patients included, there were recurrences in both groups, raising questions about the relevance of the study.
  * One serious complication in one group was reported.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOI/2020/2021/JF-01
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Thermoablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Procedure: Thermoablation with standard CT guidance
- Porto-scanner guidance with Angio-CT (Experimental)
  Interventions: Procedure: Thermoablation with porto-scanner guidance with Angio-CT

INTERVENTIONS:
Procedure: Thermoablation with standard CT guidance — Guidance with small volume breathing and high frequency. The contrast product will be venously injected in the elbow.
  Arms: Control
Procedure: Thermoablation with porto-scanner guidance with Angio-CT — Real time guidance, small volume and high frequency respiration. Contrast medium will be directly injected into the superior mesenteric artery (SMA) after puncture of the femoral artery at the inguinal fold and catheterization of the SMA.
  Arms: Porto-scanner guidance with Angio-CT

SUMMARY:
Hepatic metastases of colorectal cancer (CRC) are partially necrotic tumors mainly vascularized by the hepatic artery. When resectable, these metastases must be removed with a safety margin of 1 mm. Resection margins greater than 1 cm are associated with better disease-free survival and no local recurrence. Thermoablation systems allow for ablation zones of approximately 4.5-5 cm in diameter. For tumors <3 cm, subject to perfect targeting, it is possible to obtain ablation margins of 1 cm, which would greatly reduce the local recurrence rate. Accurate assessment of these tumor boundaries and characterization of these margins are paramount to ensure complete ablation.

Thermoablation for these small liver metastases (<3cm) has shown equivalent efficacy to surgery in terms of recurrence and survival with fewer complications. Thermoablation treatment is indicated for patients with stable disease undergoing chemotherapy. This leads to liver remodeling and metastases become difficult to see on ultrasound and CT scans. The study authors hypothesize that the porto-scanner guidance technique with Angio-CT for thermoablation treatment of CRC liver metastases will allow a better exploration of these metastases by allowing a better identification of the margins and thus ensure a more accurate and complete treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patients with CRC liver metastases (< 3 lesions, < 3 cm in diameter), proven on MRI and/or Positron Emission Tomography scan.
* Patient eligible for thermoablation requiring CT guidance (at least one metastasis not visible on ultrasound).
* Treatment by thermoablation validated in multidisciplinary meeting.
* Eastern Cooperative Oncology Group performance score 0-2.
* ASA score 1-3.
* Life expectancy of more than 3 months.
* Renal function allowing iodinated contrast injection (clearance > 30 mL/min), normal liver function (bilirubin < 35 µmol/L) and hemostasis assessment allowing percutaneous procedure (PT > 50%, platelets > 50 G/L, anticoagulant treatment to be stopped).
* Postmenopausal patient or patient with effective contraception (hormonal or mechanical)
* Pregnancy test (bHCG blood) negative in the month prior to inclusion for patients of childbearing age

  * Patients with a history of radical treatment (surgery, radiofrequency or stereotactic radiotherapy) for liver metastases more than 6 months old.
  * Patient presenting a recurrence at a distance from the treated lesion (more than 1 cm from the scar).

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Lesion not eligible for thermoablation (proximity of the liver hilum and the main bile duct).
* Uncorrectable abnormalities of liver or blood functions (coagulation).
* Severe allergy to contrast media.
* Contraindication to MRI (pacemaker, neuro-stimulator, cochlear implant, metallic heart valve, claustrophobia).
* Uncontrolled infection.
* Any physical, physiological or psychological condition incompatible with study participation or patient compliance.
* Pregnant, parturient or nursing patient.
* Contraindications mentioned in the Product Monographs of the following drugs:

  * FLUCIS: Hypersensitivity to the active substance (fludeoxyglucose (18F)) or to one of the excipients.
  * VISIPAQUE 320
  * Hypersensitivity to the active substance or to any of the excipients mentioned in section 6.1.
  * History of immediate major or delayed cutaneous reaction (see section 4.8) to the injection of iodinated contrast material (Visipaque),
  * Decompensated cardiac insufficiency with systemic injection (only concerns high osmolarity ionic products),
  * Overt thyreotoxicosis,
  * Hysterosalpingography in pregnancy

    * patient with a history of radical treatment for liver metastases (surgery, thermoablation, stereotactic radiotherapy) less than 6 months old.
    * patient with recurrence within 1 cm of the scar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of conventional CT versus porto-scanner for thermoablation of colorectal cancer liver metastases between groups | 3 months
  Percentage, where complete response is defined as complete ablation of the treated lesions (complete disappearance of enhancement and hypermetabolism) with no new lesions appearing, determined on imaging.

SECONDARY OUTCOMES:
Difference in response rate per lesion between the groups | 3 months
  Percentage
Difference in distant recurrences between the groups | 12 Months
Difference in local recurrences between the groups | 12 Months
  Yes/no presence of recurrence
Recurrence free survival between the groups | 12 months
  Days
Local recurrence-free survival between the groups | 12 months
  Days
Distant recurrence-free survival between the groups | 12 months
  Days
Difference in time until recurrence between the groups | 12 months
  Days
Size of the lesions | 3 months
  mm
Diameter of the tumor in axial | 3 months
  mm
Location of the lesions | 3 months
  Dome/left liver/sub capsular/contact with a large vessel (> 5mm)
Size of the ablation area | 3 months
  mm
Feasibility of porto-scanner | End of procedure (Day 0)
  Presence of metastatic lesions by scanner yes/no
Complications arising during intervention | End of procedure (Day 0) until 3 months
  Complications related to the approach (vascular complications), related to the percutaneous procedure (hematoma, active bleeding) or related to the treatment; Clavien-Dindo classification
Reason for for failure of technique requiring switch to different guidance technique | End of procedure (Day 0)
  Vascular problem (failure of catheterization) or problem of elevation (no optimal elevation of the liver allowing guidance)
Cost estimates for both guidance techniques during intervention | End of procedure (Day 0)
  Cost differential of the two guidance techniques for thermoablation of colorectal cancer liver metastases from the point of view of the healthcare facility

CONTACTS AND LOCATIONS:
Overall Officials: Julien Frandon, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

REFERENCES:
- [Result] Doppelt G, de Oliviera F, Minier C, Chevallier T, Beregi JP, Guiu B, Frandon J. MARGIN: Randomized Trial of Arterial CT Portography Versus Standard Imaging Guidance for Percutaneous Thermal Ablation of Colorectal Liver Metastases. Cardiovasc Intervent Radiol. 2025 Dec 28. doi: 10.1007/s00270-025-04267-5. Online ahead of print. PMID 41457158